CLINICAL TRIAL: NCT04876404
Title: Somatotopy and Striatal Plasticity in Parkinson's Disease
Brief Title: Somatotopy in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Pacific Parkinson's Research Centre (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, A. Jon Stoessl, Professor & Head of Neurology, Pacific Parkinson's Research Centre
Other Study IDs: H19-03166
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Positron-Emission Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Parkinson's Disease: Individuals with early stage Parkinson's Disease (diagnosed within the last 5 years)
  Interventions: Diagnostic Test: PET/MR Imaging
- Healthy Controls: Healthy control individuals with no neurological or mood disorders.
  Interventions: Diagnostic Test: PET/MR Imaging

INTERVENTIONS:
Diagnostic Test: PET/MR Imaging — The hybrid PET/MR scanner can provide information on brain activity during various motor and cognitive tasks.
  Other Names: Positron Emission Tomography and Magnetic Resonance Imaging

SUMMARY:
This study aims to assess changes in connections within the brain in Parkinson's disease (PD). We will invite up to 10 people with PD to participate in this study and complete several brain scans using PET (Positron Emission Tomography) and fMRI (functional Magnetic Resonance Imaging) on the Hybrid PET/MRI scanner. We will also invite 10 participants without PD to complete the same scans for comparison. "Somatotopy" refers to how areas of the brain are organized according to the body part they affect. The striatum is the brain region that coordinates complex thinking and movement. Plasticity refers to changes in connections within the brain, which can happen to make up for changes that are related to PD. In this study we will use PET and fMRI imaging together to investigate changes in the striatum in people affected by Parkinson's disease. The hybrid PET/MR scanner allows us to perform simultaneous PET and MRI measurements to investigate this.

DETAILED DESCRIPTION:
Purpose

The current investigation aims to study the altered striatal plasticity in early stage PD versus healthy controls to delineate the functional reorganization of dopaminergic projections in PD neurodegeneration. Analysis will be initially restricted to early PD, when compensatory mechanisms are likely compensating for deficits arising from dopamine deficiency. The use of hybrid PET-MRI imaging will allow for the simultaneous assessment of patterns of striatal activation and functional connectivity, as well as dopamine release induced by a variety of cognitive and motor tasks. In the future, depending upon the findings of this study, we will examine the effects of disease progression on segregation of striatal function. Altered plasticity is likely to contribute to clinical progression of disease and to disease and treatment related complications, thus this investigation may help advance the development of more effective PD treatment measures.

This investigation is intended as a pilot study. We currently do not have data on which to base a power analysis for sample size, however based on our previous experience using a double or triple bolus [11C] raclopride techniques, a sample size of 10 individuals per study group is adequate to detect between-group differences in dopamine release using a single bolus technique. Previous investigations we will be referencing in our study have similarly relied on small sample sizes to obtain their data.

We are specifically interested in tracking functional changes within the brain in early PD, as this is when compensatory mechanisms are still compensating for deficits arising from dopamine deficiency. Thus for the purposes of this investigation we would like to focus on early PD, with the potential to follow the PD cohort in a longitudinal fashion in future investigations, to assess progressive loss of segregation over time.

Hypotheses

1. In healthy subjects, there will be segregation of striatal activation as measured by cerebral blood flow determined by BOLD fMRI, as well as striatal dopamine release determined using simultaneous [11C]raclopride PET, according to body site (motor activation) and task type (motor vs. cognitive vs. reward)
2. In patients with PD, this segregation will be lost in a progressive fashion, in which caudal and dorsal striatal activation and dopamine release are lost first, with these functions shifted to progressively more rostral and ventral regions of the striatum.

Research Design

This is a cross-sectional study on 20 subjects (10 healthy control, 10 PD), involving 2-3 visits per subject to the Pacific Parkinson's Research Centre in UBC, Vancouver, BC. Each study participant will undergo 4 separate scans, 2 scans per day.

ELIGIBILITY:
Parkinson's Disease Individuals

Inclusion Criteria:

i. Recently diagnosed with early stage Parkinson's Disease (within 5 years of diagnosis) ii. Between the ages of 50 to 85 iii. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study

Healthy Control Individuals

Inclusion Criteria:

i. Healthy male between the ages of 50 and 85 ii. Healthy female between the ages of 50 and 85 iii. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study

Exclusion Criteria (All Individuals):

i. Current or past major psychiatric disorders (e.g. depression, anxiety disorders) or other major neurological disease ii. Current or past substance use problems iii. Serious head injury with loss of consciousness for ≥ 5 minutes iv. Fear of enclosed, confined spaces v. Pregnant or breastfeeding vi. Presence of active, recent, or repeated cancer vii. Unstable/undiagnosed medical conditions viii. Certain medications or conditions may impact the ability to participate and these will be discussed on a case by case basis with the study team.

ix. Weight of more 158 kg x. Inability to remain still during the scans. xi. People for whom MRI is contra-indicated:

* People with a non-MRI safe intrauterine device (IUD);
* Machinist or Metalworkers;
* Cardiac pacemaker, wires or defibrillator;
* Past injury where a piece of metal lodged in your eye or orbit;
* Ferromagnetic aneurysm clip;
* Artificial heart valve;
* Brain aneurysm clip;
* Electrical stimulator for nerves or bones or brains;
* Ear or eye implant;
* Implanted drug infusion pump;
* Coil, catheter, or filter in any blood vessel;
* Orthopaedic hardware (artificial joint, plate, screws);
* Other metallic prostheses;
* Shrapnel, bullets, or other metal fragments;
* Surgery (brain or otherwise), tattoos or injection into a join in the last 6 weeks

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with Parkinson's Disease and those without.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Striatal Dopamine Release | Baseline
  [11C]raclopride PET
Striatal Activation | Baseline
  BOLD fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Jess McKenzie, Study Director — Pacific Parkinson's Research Centre
Locations (1):
- UBC Pacific Parkinson's Research Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No